## The Effects of the Pilates Method on Pelvic Floor Injuries during Pregnancy and Childbirth: A Quasi-experimental Study

| NC | т | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| INC | • | • | • • | • | • | • | • | • | • | • | • | • | • | • | • | • | • | • | • | • | • | • | • | • | • | • | - | • | • | • | • | • | • | • | • |

Data: 10/10/2018

## PATIENT INFORMATION ABOUT THE STUDY

TITLE: Impact of The Pilates Method on Pelvic Floor Injuries During Pregnancy.

We propose you to participate in a study that will be carried out in your health centre about the injuries of the floor during childbirth. Your participation is very important because you will be helping to improve the health of many other pregnant women.

For this purpose, between the eighth and tenth day after giving birth, you will be given a telephone survey about the evolution of the study.

Your personal data will be collected in complete confidentiality, and the research team will be responsible for it. Confidentiality will always be maintained with regard to any information you give us.

Throughout the study we will always be available to answer any questions or doubts you may have.

Your participation will always be voluntary and if at any time you wish to leave the study, this will never influence the treatment of you or your health.

Thank you very much for your participation.

## PATIENT'S INFORMED CONSENT

I declare that:

- I have read and understood the information sheet given to me about the study.
- I have been able to ask questions about the study and my doubts have been clarified.
  - I have received information about the study in sufficient quantity and quality.
- I understand that the data collected will be completely confidential. Professional secrecy will always be maintained.
- I understand that my participation is voluntary and that I can withdraw from the study at any time without this affecting my medical care.

For all the above reasons, I freely accept and give my consent to participate in the study.

| Signature: | ••• |
|---------------------|-----|
| Data:/201. | |
| Identification code | |